CLINICAL TRIAL: NCT00363870
Title: A Study to Demonstrate the Efficacy of GSK Biologicals' Influenza Vaccine (Fluarix™) Administered Intramuscularly in Adults
Brief Title: A Study to Demonstrate the Efficacy of GSK Biologicals' Influenza Vaccine in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 108134
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Influenza vaccine; Prophylaxis Influenza vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Fluarix vaccine

SUMMARY:
The purpose of this study is to demonstrate the efficacy of GSK Biologicals' influenza vaccine (Fluarix™) administered intramuscularly in adults.

ELIGIBILITY:
Inclusion Criteria:

* A male or female age between 18 and 64 years at the time of the first vaccination.
* non-childbearing female

Exclusion Criteria:

* Use of non-registered products
* Pregnancy
* Hypersensitivity to a previous dose of influenza vaccine
* Acute disease at the time of enrolment/vaccination.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine
* Administration of any other influenza vaccine for the season 2006-2007
* Chronic disorders of the pulmonary or cardiovascular system, including asthma.
* Administration of immune-modifying drugs
* Administration of immunoglobulins and/or any blood products
* History of requiring regular medical follow-up or hospitalization during the preceding year because of chronic metabolic diseases (including diabetes mellitus), renal dysfunction, hemoglobinopathies, asthma or immunosuppression (including immunosuppression caused by medications or by human immunodeficiency virus)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7632
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
occurrence of confirmed influenza

SECONDARY OUTCOMES:
occurrence of influenza like illness
Occurrence of pneumonia
Immune response at days 0 and 21
Safety during 7 Months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- GSK Investigational Site, Hradec Králové, Czechia
- Finland (12):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vesikari T, Beran J, Durviaux S, Stainier I, El Idrissi M, Walravens K, Devaster JM. Use of real-time polymerase chain reaction (rtPCR) as a diagnostic tool for influenza infection in a vaccine efficacy trial. J Clin Virol. 2012 Jan;53(1):22-8. doi: 10.1016/j.jcv.2011.10.013. Epub 2011 Nov 11. PMID 22079305
- [Derived] Beran J, Vesikari T, Wertzova V, Karvonen A, Honegr K, Lindblad N, Van Belle P, Peeters M, Innis BL, Devaster JM. Efficacy of inactivated split-virus influenza vaccine against culture-confirmed influenza in healthy adults: a prospective, randomized, placebo-controlled trial. J Infect Dis. 2009 Dec 15;200(12):1861-9. doi: 10.1086/648406. PMID 19909082
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register